CLINICAL TRIAL: NCT05611437
Title: Ultrafast Ultrasonographic Oro-laryngeal Measurement in Critically Ill Patients During Weaning From Mechanical Ventilation
Acronym: REVEAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01363-40
Record Dates: First submitted 2022-10-10; First posted 2022-11-10 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Laryngeal Edema
Keywords: Post-extubation stridor; Intensive care unit; Ultrafast ultrasonography
MeSH Terms: conditions — Laryngeal Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrafast ultrasonography — Ultrasonography of the neck, patient in supine position, neck hyper-extended. Three different scanning planes containing several landmarks. Carried out in the 12h prior extubation.

SUMMARY:
In ICU, ventilatory weaning failure is common, accounting for up to 25% of extubations. These failures are largely due to swallowing disorders and laryngeal edema. Edema prevalence in ICU varies between 4 and 37%.

Post-extubation stridor is a clinical sign of upper airway obstruction and may require urgent reintubation, which is associated with increased patient length of stay, morbidity and mortality.

Identifying patients at risk is critical, and the need for reliable tools to predict the occurence of laryngeal edema is still relevant.

ELIGIBILITY:
Inclusion Criteria:

* Adults,
* Intubated and ventilated for more than 24h,
* Filing mechanical ventilation weaning criteria.

Exclusion Criteria:

* Pregnant of breast-feeding woman,
* Under guardianship patient,
* History of laryngeal tumor, stroke, paralysis of recurrent nerve, swallowing disorders,
* History of surgical laryngeal intervention or radiotherapy,
* Unplanned extubation,
* Opposition to take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted in Le Havre Hospital intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between laryngeal ultrafast ultrasonography and occurence of laryngeal edema | Within the 24 hours following extubation
  A laryngeal edema is defined as a post-extubation stridor. Performance of ultrafast ultrasonography for laryngeal edema prediction in intensive care patients will be assessed with specificity, sensitivity, positive predictive value and negative predictive value.

SECONDARY OUTCOMES:
Correlation between laryngeal ultrafast ultrasonography and occurence of swallowing disorders | Within the 24 hours following extubation
  Performance of ultrafast ultrasonography for swallowing disorsders prediction in intensive care patients will be assessed with specificity, sensitivity, positive predictive value and negative predictive value.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier du Havre, Montivilliers, France

IPD SHARING:
Plan to Share IPD: Undecided